CLINICAL TRIAL: NCT05151744
Title: A Phase II, Multicenter, Randomized, Double Masked, Active Comparator-Controlled Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7200220 in Combination With Ranibizumab Administered Intravitreally in Patients With Diabetic Macular Edema
Brief Title: A Study to Investigate Vamikibart (RO7200220) in Combination With Ranibizumab in Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP43464; 2021-004390-31 (EudraCT Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Vamikibart + Ranibizumab (Experimental): Participants will receive vamikibart, 1 milligram (mg) administered as intravitreal (IVT) injection in combination with ranibizumab, 0.5 mg IVT, on Day 1 and every fourth week (Q4W) up to Week 44, for a total of 12 injections, followed by an observational period up to Week 72.
  Interventions: Drug: Vamikibart; Drug: Ranibizumab
- Arm B: Ranibizumab (Active Comparator): Participants will receive ranibizumab, 0.5 mg IVT, from Day 1 and Q4W in combination with sham up to Week 44, for a total of 12 injections, followed by an observational period up to Week 72.
  Interventions: Drug: Ranibizumab; Other: Sham Procedure

INTERVENTIONS:
Drug: Vamikibart — Vamikibart will be administered by IVT injection in the study eye.
  Other Names: RO7200220
  Arms: Arm A: Vamikibart + Ranibizumab
Drug: Ranibizumab — Ranibizumab will be administered by IVT injection in the study eye.
  Other Names: Lucentis
Other: Sham Procedure — Sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye.
  Arms: Arm B: Ranibizumab

SUMMARY:
Study BP43464 is a phase II, multicenter, randomized, double-masked active comparator-controlled study designed to assess the efficacy, safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of vamikibart in combination with, anti-vascular endothelial growth factor (VEGF) inhibitor, ranibizumab compared with ranibizumab alone in participants with diabetic macular edema. Only one eye will be chosen as the study eye. The duration of the study will be 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (Type 1 or Type 2)
* Macular thickening secondary to diabetic macular edema (DME) involving the center of the macula
* Decreased visual acuity attributable primarily to DME
* Ability and willingness to provide written informed consent and to comply with the study protocol
* Willingness to allow Aqueous Humor collection
* For women of childbearing potential: agreement to remain abstinent or use at least one highly effective contraceptive method that results in a failure rate of <1% per year during the treatment period and for at least 12 weeks after the final dose of study treatment

Exclusion Criteria:

* Hemoglobin A1c (HbA1c) of greater than (>) 12%
* Uncontrolled blood pressure, defined as a systolic value greater than (>)180 millimeters of mercury (mmHg) and/or a diastolic value >100 mmHg while a patient is at rest
* Currently pregnant or breastfeeding, or intend to become pregnant during the study
* Prior treatment with panretinal photocoagulation or macular laser to the study eye
* Any intraocular or periocular corticosteroid treatment within the past 16 weeks prior to Day 1 to the study eye
* Prior Iluvien or Retisert implants within 3 years prior to Day 1 to the study eye
* Prior or concomitant treatment with anti-VEGF therapy within 8 weeks prior to Day 1 to the study eye; Vabysmo^TM within 16 weeks prior to Day 1, prior Beovu® is not permitted
* Prior administration of IVT brolucizumab (Beovu®): ever; vamikibart: </=24 weeks prior to Day 1) in either eye
* Any proliferative diabetic retinopathy
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye
* Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (10):
  - Win Retina, Arcadia, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Florida Eye Associates, Melbourne, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Deep Blue Retina PLLC, Southaven, Mississippi
  - Verum Research LLC, Eugene, Oregon
  - Texas Retina Associates, Arlington, Texas
  - Retina Consultants of Texas, Bellaire, Texas
- Argentina (5):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Centro Oftalmológico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Grupo Laser Vision, Rosario
- Canada (3):
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
- Poland (4):
  - Niepubliczny Zak?ad Opieki Zdrowotnej PRYZMAT-OKULISTYKA, Gliwice
  - Centrum Medyczne UNO-MED, Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - Caminomed, Tarnowskie Góry
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (2):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Clinica Universitaria de Navarra, Madrid
- United Kingdom (3):
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Royal Surrey County Hospital, Guildford
  - Kings College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 187 participants with diabetic macular edema (DME) took part in the study at 37 investigative sites across the United States, Argentina, Israel, South Korea, Poland, Canada, Spain, and the United Kingdom from 17 December 2021 to 1 October 2024.
Pre-assignment Details: Participants were randomized in 1:1 ratio to Vamikibart + Ranibizumab arm and Ranibizumab arm.
Groups:
- Arm A: Vamikibart + Ranibizumab: Participants received vamikibart, 1 milligrams (mg) as intravitreal (IVT) injection, every 4 weeks (Q4W) in combination with ranibizumab, 0.5 mg as IVT injection, Q4W up to Week 44 followed by an observational period up to Week 72.
- Arm B: Ranibizumab: Participants received ranibizumab, 0.5 mg as an IVT injection, Q4W in combination with sham treatment up to Week 44 followed by an observational period up to Week 72.
Period: Overall Study
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Started | 93 | 94
Previously-treated Intent-to-treat (ITT) Population (Previously-treated ITT population included all randomized participants who were IVT anti-vascular endothelial growth factor (anti-VEGF) or periocular/IVT corticosteroids previously treated participants as defined in the exclusion criteria 9 and 10 in the protocol.) | 32 | 31
Treatment-naive ITT Population (Treatment-naïve ITT population included all randomized participants who were IVT anti-VEGF or periocular/IVT corticosteroids treatment-naïve as defined in the exclusion criteria 9 and 10 in the protocol.) | 61 | 63
Completed | 64 | 81
Not Completed | 29 | 13
Not completed — Adverse Event | 6 | 2
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Need for Rescue Treatment | 0 | 1
Not completed — Non-compliance with Study Drug | 0 | 1
Not completed — Reason not Specified | 10 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Population: ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Groups:
- Arm A: Vamikibart + Ranibizumab: Participants received vamikibart, 1 mg as IVT injection, Q4W in combination with ranibizumab, 0.5 mg as IVT injection, Q4W up to Week 44 followed by an observational period up to Week 72.
- Total: Total of all reporting groups
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.1) | 62.1 (9.3) | 61.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 62 | 55 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 14 | 20
  Not Hispanic or Latino | 56 | 56 | 112
  Unknown or Not Reported | 31 | 24 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 45 | 60 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 31 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Averaged Over Week 44 and Week 48 in Treatment-naïve Participants
Description: BCVA was measured via Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters using a set of three Precision vision^TM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity (VA) examiner. The BCVA letter score ranges from 0 to 100 letters. Higher scores and gain in BCVA from baseline indicate improvement in VA. This analysis used a Mixed Model for Repeated Measurements (MMRM) model.
Time Frame: Baseline, Week 44 and Week 48
Population: Treatment naïve ITT population included all randomized participants who were IVT anti-vascular endothelial growth factor (anti-VEGF) or periocular/IVT corticosteroids treatment-naïve as defined in the exclusion criteria 9 and 10 in the protocol.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
letters | 12.8 (1.30) | 9.4 (1.25)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.0625, MMRM; Difference in Adjusted Means = 3.4, 95% CI 2-sided [-0.2 to 7.0]

2. Secondary Outcome: Number of Participants With Systemic and Ocular Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Systemic AEs include all non-ocular AEs.
Time Frame: Up to Week 72
Population: Safety Population included all participants randomized to study treatment and received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
Participants
  Systemic AEs | 54 | 60
  Ocular AEs in Study Eyes | 33 | 28
  Ocular AEs in Fellow Eyes | 25 | 27

3. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 44 and Week 48 in Previously Treated Participants
Description: BCVA was measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision vision^TM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The BCVA letter score ranges from 0 to 100 letters. Higher scores and gain in BCVA from baseline indicate improvement in VA. This analysis used a MMRM model.
Time Frame: Baseline, Week 44 and Week 48
Population: Previously treated ITT population included all randomized participants who were IVT anti-VEGF or periocular/IVT corticosteroids previously treated participants as defined in the exclusion criteria 9 and 10 in the protocol.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
letters | 11.1 (1.50) | 8.4 (1.49)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.2052, MMRM; Difference in Adjusted Mean = 2.7, 95% CI 2-sided [-1.5 to 7.0]

4. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 44 and Week 48 in Overall ITT Population
Description: as for outcome 3
Time Frame: Baseline, Week 44 and Week 48
Population: Overall ITT population included all randomized participants grouped according to the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
letters | 12.4 (0.99) | 9.1 (0.96)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.0192, MMRM; Difference in Adjusted Mean = 3.3, 95% CI 2-sided [0.5 to 6.0]

5. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Treatment-naïve Participants
Description: as for outcome 3
Time Frame: Baseline, Week 32 and Week 36
Population: Treatment-naïve ITT population included all randomized participants who were IVT anti-VEGF or periocular/IVT corticosteroids treatment-naïve as defined in the exclusion criteria 9 and 10 in the protocol.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
letters | 11.8 (0.97) | 9.3 (0.94)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.0637, MMRM; Difference in Adjusted Mean = 2.5, 95% CI 2-sided [-0.1 to 5.2]

6. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Previously Treated Participants
Description: as for outcome 3
Time Frame: Baseline, Week 32 and Week 36
Population: as for outcome 3
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
letters | 8.3 (1.43) | 7.5 (1.46)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.7091, MMRM; Difference in Adjusted Mean = 0.8, 95% CI 2-sided [-3.3 to 4.9]

7. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 32 and Week 36, in Overall ITT Population
Description: as for outcome 3
Time Frame: Baseline, Week 32 and Week 36
Population: as for outcome 4
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
letters | 10.6 (0.81) | 8.7 (0.80)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.1107, MMRM; Difference in Adjusted Mean = 1.8, 95% CI 2-sided [-0.4 to 4.1]

8. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 20 and Week 24 in Treatment-naïve Participants
Description: as for outcome 3
Time Frame: Baseline, Week 20 and Week 24
Population: Treatment naïve ITT population included all randomized participants who were IVT anti-VEGF or periocular/IVT corticosteroids treatment-naïve as defined in the exclusion criteria 9 and 10 in the protocol.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
letters | 10.6 (1.04) | 8.5 (1.01)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.1498, MMRM; Difference in Adjusted Mean = 2.1, 95% CI 2-sided [-0.8 to 5.0]

9. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 20 and Week 24 in Previously Treated Participants
Description: as for outcome 3
Time Frame: Baseline, Week 20 and Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
letters | 8.1 (1.46) | 6.2 (1.47)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.3783, MMRM; Difference in Adjusted Mean = 1.8, 95% CI 2-sided [-2.3 to 6.0]

10. Secondary Outcome: Change From Baseline in BCVA Averaged Over Week 20 and Week 24, in Overall ITT Population
Description: as for outcome 3
Time Frame: Baseline, Week 20 and Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
letters | 9.7 (0.84) | 7.8 (0.83)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.1036, MMRM; Difference in Adjusted Mean = 1.9, 95% CI 2-sided [-0.4 to 4.3]

11. Secondary Outcome: Change From Baseline in BCVA Over Time in Overall ITT Population
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: Overall ITT population included all randomized participants grouped according to the treatment assigned at randomization. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
letters
  Baseline | 62.6 (1.02) | 62.0 (1.01)
  Change at Week 4: number analyzed (Participants) | 92 | 90
  Change at Week 4 | 6.7 (0.64) | 4.2 (0.65)
  Change at Week 8: number analyzed (Participants) | 88 | 90
  Change at Week 8 | 7.6 (0.76) | 4.6 (0.76)
  Change at Week 12: number analyzed (Participants) | 89 | 92
  Change at Week 12 | 8.9 (0.78) | 6.4 (0.78)
  Change at Week 16: number analyzed (Participants) | 89 | 87
  Change at Week 16 | 9.3 (0.83) | 7.4 (0.83)
  Change at Week 20: number analyzed (Participants) | 83 | 91
  Change at Week 20 | 9.7 (0.81) | 7.6 (0.80)
  Change at Week 24: number analyzed (Participants) | 85 | 86
  Change at Week 24 | 9.8 (1.03) | 8.0 (1.02)
  Change at Week 28: number analyzed (Participants) | 85 | 87
  Change at Week 28 | 10.1 (0.87) | 8.5 (0.87)
  Change at Week 32: number analyzed (Participants) | 80 | 80
  Change at Week 32 | 10.5 (0.88) | 8.8 (0.87)
  Change at Week 36: number analyzed (Participants) | 73 | 83
  Change at Week 36 | 10.6 (0.84) | 8.6 (0.83)
  Change at Week 40: number analyzed (Participants) | 74 | 85
  Change at Week 40 | 10.9 (0.95) | 8.8 (0.93)
  Change at Week 44: number analyzed (Participants) | 67 | 79
  Change at Week 44 | 12.2 (1.01) | 8.7 (0.99)
  Change at Week 48: number analyzed (Participants) | 68 | 81
  Change at Week 48 | 12.5 (1.03) | 9.4 (1.00)
  Change at Week 52: number analyzed (Participants) | 70 | 81
  Change at Week 52 | 11.1 (1.07) | 8.0 (1.03)
  Change at Week 56: number analyzed (Participants) | 67 | 75
  Change at Week 56 | 10.8 (1.13) | 7.8 (1.09)
  Change at Week 60: number analyzed (Participants) | 61 | 64
  Change at Week 60 | 10.4 (1.18) | 7.7 (1.14)
  Change at Week 64: number analyzed (Participants) | 57 | 53
  Change at Week 64 | 10.2 (1.12) | 8.2 (1.10)
  Change at Week 68: number analyzed (Participants) | 53 | 49
  Change at Week 68 | 9.9 (1.14) | 7.6 (1.11)
  Change at Week 72: number analyzed (Participants) | 52 | 45
  Change at Week 72 | 9.2 (1.12) | 7.8 (1.11)

12. Secondary Outcome: Percentage of Participants Gaining ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA Over Time in Overall ITT Population
Description: BCVA was measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision vision^TM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The BCVA letter score ranges from 0 to 100 letters. Higher scores indicate improvement in VA. Percentages have been rounded off.
Time Frame: Up to Week 72
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Participants Gaining ≥ 0 Letters | 98.9 | 98.9
  Participants Gaining ≥ 5 Letters | 94.6 | 90.4
  Participants Gaining ≥ 10 Letters | 76.3 | 69.1
  Participants Gaining ≥ 15 Letters | 49.5 | 44.7

13. Secondary Outcome: Percentage of Participants Losing ≥ 15, ≥ 10, or ≥ 5 Letters in BCVA Over Time in Overall ITT Population
Description: as for outcome 12
Time Frame: Up to Week 72
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Participants Losing ≥ 5 Letters | 19.4 | 27.7
  Participants Losing ≥ 10 Letters | 7.5 | 11.7
  Participants Losing ≥ 15 Letters | 4.3 | 6.4

14. Secondary Outcome: Percentage of Participants With BCVA ≥ 69 Letters (20/40 Snellen Equivalent) Over Time
Description: BCVA was measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision vision^TM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The BCVA letter score ranges from 0 (Snellen equivalent <20/800) to 100 (Snellen equivalent of 20/10) letters. Higher scores indicate improvement in VA. Percentages have been rounded off.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline | 34.4 | 31.9
  Week 1: number analyzed (Participants) | 88 | 90
  Week 1 | 53.4 | 48.9
  Week 4: number analyzed (Participants) | 92 | 90
  Week 4 | 63.0 | 53.3
  Week 8: number analyzed (Participants) | 88 | 90
  Week 8 | 67.0 | 48.9
  Week 12: number analyzed (Participants) | 89 | 92
  Week 12 | 73.0 | 56.5
  Week 16: number analyzed (Participants) | 89 | 87
  Week 16 | 69.7 | 57.5
  Week 20: number analyzed (Participants) | 83 | 91
  Week 20 | 74.7 | 67.0
  Week 24: number analyzed (Participants) | 85 | 86
  Week 24 | 70.6 | 61.6
  Week 28: number analyzed (Participants) | 85 | 87
  Week 28 | 71.8 | 63.2
  Week 32: number analyzed (Participants) | 80 | 80
  Week 32 | 78.8 | 62.5
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 72.6 | 62.7
  Week 40: number analyzed (Participants) | 74 | 85
  Week 40 | 78.4 | 70.6
  Week 44: number analyzed (Participants) | 67 | 79
  Week 44 | 82.1 | 67.1
  Week 48: number analyzed (Participants) | 68 | 81
  Week 48 | 80.9 | 70.4
  Week 52: number analyzed (Participants) | 70 | 81
  Week 52 | 78.6 | 64.2
  Week 56: number analyzed (Participants) | 67 | 75
  Week 56 | 82.1 | 58.7
  Week 60: number analyzed (Participants) | 61 | 64
  Week 60 | 82.0 | 68.8
  Week 64: number analyzed (Participants) | 57 | 53
  Week 64 | 82.5 | 69.8
  Week 68: number analyzed (Participants) | 53 | 49
  Week 68 | 81.1 | 71.4
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 82.7 | 71.1

15. Secondary Outcome: Percentage of Participants With BCVA ≥ 84 Letters (20/20 Snellen Equivalent) Over Time
Description: as for outcome 14
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline | 0 | 0
  Week 1: number analyzed (Participants) | 88 | 90
  Week 1 | 2.3 | 0
  Week 4: number analyzed (Participants) | 92 | 90
  Week 4 | 6.5 | 2.2
  Week 8: number analyzed (Participants) | 88 | 90
  Week 8 | 10.2 | 5.6
  Week 12: number analyzed (Participants) | 89 | 92
  Week 12 | 10.1 | 8.7
  Week 16: number analyzed (Participants) | 89 | 87
  Week 16 | 13.5 | 6.9
  Week 20: number analyzed (Participants) | 83 | 91
  Week 20 | 14.5 | 8.8
  Week 24: number analyzed (Participants) | 85 | 86
  Week 24 | 17.6 | 8.1
  Week 28: number analyzed (Participants) | 85 | 87
  Week 28 | 12.9 | 11.5
  Week 32: number analyzed (Participants) | 80 | 80
  Week 32 | 17.5 | 13.8
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 13.7 | 12.0
  Week 40: number analyzed (Participants) | 74 | 85
  Week 40 | 12.2 | 11.8
  Week 44: number analyzed (Participants) | 67 | 79
  Week 44 | 23.9 | 8.9
  Week 48: number analyzed (Participants) | 68 | 81
  Week 48 | 23.5 | 14.8
  Week 52: number analyzed (Participants) | 70 | 81
  Week 52 | 15.7 | 7.4
  Week 56: number analyzed (Participants) | 67 | 75
  Week 56 | 14.9 | 9.3
  Week 60: number analyzed (Participants) | 61 | 64
  Week 60 | 13.1 | 9.4
  Week 64: number analyzed (Participants) | 57 | 53
  Week 64 | 19.3 | 11.3
  Week 68: number analyzed (Participants) | 53 | 49
  Week 68 | 18.9 | 10.2
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 11.5 | 11.1

16. Secondary Outcome: Percentage of Participants With BCVA ≤ 38 Letters (20/200 Snellen Equivalent) Over Time
Description: as for outcome 14
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline | 3.2 | 4.3
  Week 1: number analyzed (Participants) | 88 | 90
  Week 1 | 2.3 | 2.2
  Week 4: number analyzed (Participants) | 92 | 90
  Week 4 | 2.2 | 3.3
  Week 8: number analyzed (Participants) | 88 | 90
  Week 8 | 2.3 | 3.3
  Week 12: number analyzed (Participants) | 89 | 92
  Week 12 | 2.2 | 2.2
  Week 16: number analyzed (Participants) | 89 | 87
  Week 16 | 1.1 | 1.1
  Week 20: number analyzed (Participants) | 83 | 91
  Week 20 | 1.2 | 2.2
  Week 24: number analyzed (Participants) | 85 | 86
  Week 24 | 2.4 | 1.2
  Week 28: number analyzed (Participants) | 85 | 87
  Week 28 | 3.5 | 2.3
  Week 32: number analyzed (Participants) | 80 | 80
  Week 32 | 2.5 | 1.3
  Week 36: number analyzed (Participants) | 73 | 83
  Week 36 | 1.4 | 1.2
  Week 40: number analyzed (Participants) | 74 | 85
  Week 40 | 2.7 | 2.4
  Week 44: number analyzed (Participants) | 67 | 79
  Week 44 | 1.5 | 1.3
  Week 48: number analyzed (Participants) | 68 | 81
  Week 48 | 0 | 1.2
  Week 52: number analyzed (Participants) | 70 | 81
  Week 52 | 1.4 | 0
  Week 56: number analyzed (Participants) | 67 | 75
  Week 56 | 3.0 | 0
  Week 60: number analyzed (Participants) | 61 | 64
  Week 60 | 1.6 | 1.6
  Week 64: number analyzed (Participants) | 57 | 53
  Week 64 | 1.8 | 0
  Week 68: number analyzed (Participants) | 53 | 49
  Week 68 | 1.9 | 0
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 0 | 0

17. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST) Averaged Over Week 44 and Week 48 in Treatment-naïve Participants
Description: CST was defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield. CST was measured using spectral domain optical coherence tomography (SD-OCT). Negative change from baseline values denotes improvement. This analysis used a MMRM model.
Time Frame: Baseline, Week 44 and Week 48
Population: as for outcome 8
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
μm | -202.4 (10.63) | -192.4 (10.11)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.4968, MMRM; Difference in Adjusted Mean = -10.0, 95% CI 2-sided [-38.9 to 18.9]

18. Secondary Outcome: Change From Baseline in CST Averaged Over Week 44 and Week 48 in Previously Treated Participants
Description: CST was defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 mm central subfield. CST was measured using SD-OCT. Negative change from baseline values denotes improvement. This analysis used a MMRM model.
Time Frame: Baseline, Week 44 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: micrometre (μm)
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
micrometre (μm) | -194.4 (19.58) | -171.2 (18.79)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.3951, MMRM; Difference in Adjusted Mean = -23.2, 95% CI 2-sided [-76.8 to 30.5]

19. Secondary Outcome: Change From Baseline in CST Averaged Over Week 44 and Week 48 in Overall ITT Population
Description: CST was defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 mm central subfield. CST was measured using SD-OCT. Negative change from baseline values denotes improvement. This analysis used an MMRM model.
Time Frame: Baseline, Week 44 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
μm | -201.6 (8.33) | -178.8 (8.15)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.0521, MMRM; Difference in Adjusted Mean = -22.8, 95% CI 2-sided [-45.8 to 0.2]

20. Secondary Outcome: Change From Baseline in CST Averaged Over Week 32 and Week 36 in Treatment-naïve Participants
Description: as for outcome 19
Time Frame: Baseline, Week 32 and Week 36
Population: as for outcome 8
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
μm | -197.9 (10.26) | -180.3 (9.97)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.2227, MMRM; Difference in Adjusted Mean = -17.5, 95% CI 2-sided [-45.7 to 10.7]

21. Secondary Outcome: Change From Baseline in CST Averaged Over Week 32 and Week 36 in Previously Treated Participants
Description: as for outcome 19
Time Frame: Baseline, Week 32 and Week 36
Population: as for outcome 3
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
μm | -177.2 (18.38) | -150.0 (18.38)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.2972, MMRM; Difference in Adjusted Mean = -27.2, 95% CI 2-sided [-78.6 to 24.2]

22. Secondary Outcome: Change From Baseline Averaged Over Week 32 and Week 36 in Overall ITT Population
Description: as for outcome 19
Time Frame: Baseline, Week 32 and Week 36
Population: as for outcome 4
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
μm | -191.4 (8.51) | -172.1 (8.38)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.1071, MMRM; Difference in Adjusted Mean = -19.4, 95% CI 2-sided [-42.9 to 4.2]

23. Secondary Outcome: Change From Baseline in CST Averaged Over Week 20 and Week 24 in Treatment-naïve Participants
Description: as for outcome 19
Time Frame: Baseline, Week 20 and Week 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 61 | 63
μm | -184.3 (10.05) | -169.7 (9.89)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.3030, MMRM; Difference in Adjusted Mean = -14.6, 95% CI 2-sided [-42.4 to 13.2]

24. Secondary Outcome: Change From Baseline in CST Averaged Over Week 20 and Week 24 in Previously Treated Participants
Description: as for outcome 19
Time Frame: Baseline, Week 20 and Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 32 | 31
μm | -163.2 (17.75) | -120.2 (17.65)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.0878, MMRM; Difference in Adjusted Mean = -43.0, 95% CI 2-sided [-92.4 to 6.4]

25. Secondary Outcome: Change From Baseline in CST Averaged Over Week 20 and Week 24 in Overall ITT Population
Description: as for outcome 19
Time Frame: Baseline, Week 20 and Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
μm | -176.1 (9.89) | -153.9 (9.80)
Statistical Analysis 1: Comparison: Arm A: Vamikibart + Ranibizumab vs Arm B: Ranibizumab; Test type: Superiority; p = 0.1111, MMRM; Difference in Adjusted Mean = -22.3, 95% CI 2-sided [-49.8 to 5.2]

26. Secondary Outcome: Change From Baseline in CST Over Time in Overall ITT Population
Description: as for outcome 19
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 11
Measure: Mean (Standard Error); unit: μm
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
μm
  Baseline: number analyzed (Participants) | 92 | 94
  Baseline | 493.0 (11.55) | 498.4 (14.10)
  Change at Week 4: number analyzed (Participants) | 90 | 89
  Change at Week 4 | -121.0 (9.82) | -92.2 (9.77)
  Change at Week 8: number analyzed (Participants) | 86 | 90
  Change at Week 8 | -138.9 (9.67) | -108.2 (9.59)
  Change at Week 12: number analyzed (Participants) | 87 | 91
  Change at Week 12 | -147.9 (9.63) | -125.3 (9.54)
  Change at Week 16: number analyzed (Participants) | 87 | 87
  Change at Week 16 | -158.6 (10.28) | -138.3 (10.19)
  Change at Week 20: number analyzed (Participants) | 81 | 89
  Change at Week 20 | -172.8 (10.11) | -149.8 (10.00)
  Change at Week 24: number analyzed (Participants) | 85 | 86
  Change at Week 24 | -174.1 (10.12) | -152.9 (10.02)
  Change at Week 28: number analyzed (Participants) | 82 | 87
  Change at Week 28 | -181.1 (10.53) | -154.1 (10.38)
  Change at Week 32: number analyzed (Participants) | 77 | 79
  Change at Week 32 | -186.4 (8.87) | -165.6 (8.77)
  Change at Week 36: number analyzed (Participants) | 73 | 82
  Change at Week 36 | -191.1 (9.58) | -174.9 (9.33)
  Change at Week 40: number analyzed (Participants) | 75 | 84
  Change at Week 40 | -193.4 (8.92) | -166.7 (8.76)
  Change at Week 44: number analyzed (Participants) | 67 | 79
  Change at Week 44 | -197.3 (8.95) | -172.7 (8.73)
  Change at Week 48: number analyzed (Participants) | 68 | 80
  Change at Week 48 | -200.1 (9.04) | -179.2 (8.84)
  Change at Week 52: number analyzed (Participants) | 68 | 81
  Change at Week 52 | -172.7 (12.92) | -136.9 (12.25)
  Change at Week 56: number analyzed (Participants) | 68 | 75
  Change at Week 56 | -173.8 (11.43) | -129.2 (10.99)
  Change at Week 60: number analyzed (Participants) | 61 | 64
  Change at Week 60 | -155.5 (13.18) | -130.6 (12.65)
  Change at Week 64: number analyzed (Participants) | 57 | 53
  Change at Week 64 | -161.4 (13.65) | -163.0 (13.44)
  Change at Week 68: number analyzed (Participants) | 53 | 49
  Change at Week 68 | -160.1 (11.26) | -136.6 (10.96)
  Change at Week 72: number analyzed (Participants) | 52 | 45
  Change at Week 72 | -159.5 (11.62) | -154.3 (11.55)

27. Secondary Outcome: Percentage of Participants With Absence of DME Over Time in Overall ITT Population
Description: Absence of DME was defined as CST < 325 μm for Spectralis SD-OCT, or < 315 μm for Cirrus SD-OCT or Topcon SD-OCT. Percentages have been rounded off.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline: number analyzed (Participants) | 92 | 94
  Baseline | 0 [NA to NA] — The 95% CI was not estimable due to an insufficient number of participants with events. | 2.1 [0.0 to 5.0]
  Week 4: number analyzed (Participants) | 90 | 89
  Week 4 | 31.1 [21.5 to 40.7] | 25.8 [16.7 to 34.9]
  Week 8: number analyzed (Participants) | 86 | 90
  Week 8 | 45.3 [34.8 to 55.9] | 37.8 [27.8 to 47.8]
  Week 12: number analyzed (Participants) | 87 | 91
  Week 12 | 47.1 [36.6 to 57.6] | 46.2 [35.9 to 56.4]
  Week 16: number analyzed (Participants) | 87 | 87
  Week 16 | 57.5 [47.1 to 67.9] | 49.4 [38.9 to 59.9]
  Week 20: number analyzed (Participants) | 81 | 89
  Week 20 | 64.2 [53.8 to 74.6] | 60.7 [50.5 to 70.8]
  Week 24: number analyzed (Participants) | 85 | 86
  Week 24 | 65.9 [55.8 to 76.0] | 66.3 [56.3 to 76.3]
  Week 28: number analyzed (Participants) | 82 | 87
  Week 28 | 75.6 [66.3 to 84.9] | 66.7 [56.8 to 76.6]
  Week 32: number analyzed (Participants) | 77 | 79
  Week 32 | 75.3 [65.7 to 85.0] | 67.1 [56.7 to 77.5]
  Week 36: number analyzed (Participants) | 73 | 82
  Week 36 | 75.3 [65.5 to 85.2] | 73.2 [63.6 to 82.8]
  Week 40: number analyzed (Participants) | 75 | 84
  Week 40 | 77.3 [67.9 to 86.8] | 70.2 [60.5 to 80.0]
  Week 44: number analyzed (Participants) | 67 | 79
  Week 44 | 80.6 [71.1 to 90.1] | 75.9 [66.5 to 85.4]
  Week 48: number analyzed (Participants) | 68 | 80
  Week 48 | 79.4 [69.8 to 89.0] | 72.5 [62.7 to 82.3]
  Week 52: number analyzed (Participants) | 68 | 81
  Week 52 | 70.6 [59.8 to 81.4] | 55.6 [44.7 to 66.4]
  Week 56: number analyzed (Participants) | 68 | 75
  Week 56 | 67.6 [56.5 to 78.8] | 57.3 [46.1 to 68.5]
  Week 60: number analyzed (Participants) | 61 | 64
  Week 60 | 62.3 [50.1 to 74.5] | 62.5 [50.6 to 74.4]
  Week 64: number analyzed (Participants) | 57 | 53
  Week 64 | 59.6 [46.9 to 72.4] | 62.3 [49.2 to 75.3]
  Week 68: number analyzed (Participants) | 53 | 49
  Week 68 | 58.5 [45.2 to 71.8] | 61.2 [47.6 to 74.9]
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 61.5 [48.3 to 74.8] | 62.2 [48.1 to 76.4]

28. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid (IRF) Over Time in Overall ITT Population
Description: The absence of IRF in the study eye (defined as IRF absent or definite outside center subfield only) was assessed by the central reading center using SD-OCT. The percentage of participants with absence of IRF at foveal center are reported. Percentages have been rounded off.
Time Frame: Baseline, Weeks 4, 12, 24, 36, 48, and 72
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline: number analyzed (Participants) | 92 | 94
  Baseline | 19.6 | 22.3
  Week 4: number analyzed (Participants) | 89 | 90
  Week 4 | 53.9 | 47.8
  Week 12: number analyzed (Participants) | 86 | 92
  Week 12 | 60.5 | 51.1
  Week 24: number analyzed (Participants) | 82 | 86
  Week 24 | 69.5 | 69.8
  Week 36: number analyzed (Participants) | 71 | 83
  Week 36 | 70.4 | 71.1
  Week 48: number analyzed (Participants) | 66 | 78
  Week 48 | 78.8 | 78.2
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 71.2 | 75.6

29. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid (SRF) Over Time in Overall ITT Population
Description: The absence of SRF in the study eye (defined as SRF absent or definite outside center subfield only) was assessed by the central reading center using SD-OCT. The percentage of participants with absence of SRF at the foveal center are reported. Percentages have been rounded off.
Time Frame: Baseline, Weeks 4, 12, 24, 36, 48, and 72
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
Number analyzed (Participants) | 93 | 94
percentage of participants
  Baseline: number analyzed (Participants) | 91 | 94
  Baseline | 60.4 | 63.8
  Week 4: number analyzed (Participants) | 89 | 90
  Week 4 | 89.9 | 82.2
  Week 12: number analyzed (Participants) | 87 | 91
  Week 12 | 98.9 | 93.4
  Week 24: number analyzed (Participants) | 82 | 86
  Week 24 | 98.8 | 96.5
  Week 36: number analyzed (Participants) | 72 | 83
  Week 36 | 100 | 96.4
  Week 48: number analyzed (Participants) | 66 | 78
  Week 48 | 98.5 | 97.4
  Week 72: number analyzed (Participants) | 52 | 45
  Week 72 | 98.1 | 100

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: Safety population included all participants randomized to study treatment and received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
  Ocular AEs displayed include both study eye and fellow eye.
Arm/Group | Arm A: Vamikibart + Ranibizumab | Arm B: Ranibizumab
All-Cause Mortality (participants affected / at risk) | 1/93 | 2/94
Serious Adverse Events (participants affected / at risk) | 22/93 | 17/94
Other Adverse Events (participants affected / at risk) | 38/93 | 48/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Vamikibart + Ranibizumab (N=93) | Arm B: Ranibizumab (N=94)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Retinal occlusive vasculitis (Eye disorders) | 2 (2) | 0 (0)
Vitritis (Eye disorders) | 2 (2) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Vamikibart + Ranibizumab (N=93) | Arm B: Ranibizumab (N=94)
Cataract (Eye disorders) | 5 (7) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 8 (12) | 8 (8)
Diabetic retinal oedema (Eye disorders) | 9 (10) | 16 (16)
COVID-19 (Infections and infestations) | 9 (10) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 8 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypertension (Vascular disorders) | 7 (8) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT05151744/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05151744/SAP_001.pdf